CLINICAL TRIAL: NCT06656169
Title: Effect of Subcutaneous Polyvidone Collagen Treatment vs Placebo on Clinical Hand Recovery, Biochemical Response and Quality of Life in Adult Rheumatoid Arthritis.
Brief Title: Effect of Subcutaneous Polyvidone Collagen Treatment on Hand Recovery in Adult Rheumatoid Arthritis.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Polyvidone collagen effect
Record Dates: First submitted 2024-10-03; First posted 2024-10-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Collagen Polyvidone; Synovial Tissue; Tumor necrosis factor-alpha; American College of Rheumatology Questionnaire; Rheumatoid Factor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, masked, placebo-controlled, randomized clinical trial will be conducted
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Case group (Experimental): Patients with unilateral or bilateral arthritic hand, both genders, age of 60 years or older in treatment with subcutaneous polyvidone collagen.
  Interventions: Drug: Subcutaneous polyvidone collagen
- Control group (Placebo Comparator): Patients with unilateral or bilateral arthritic hand, both genders, age of 60 years or older
  Interventions: Other: saline solution

INTERVENTIONS:
Drug: Subcutaneous polyvidone collagen — Use collagen-polyvidone at a dose of 0.2 ml, applied to the affected area of the hand.
  Other Names: Fibroquel
  Arms: Case group
Other: saline solution — administer saline solution at a dose of 0.2 ml, applied to the affected area of the hand.
  Arms: Control group

SUMMARY:
A study in geriatric rheumatology on the treatment of rheumatoid arthritis (RA) in older adults is described. Its objective is to compare the effects of subcutaneous polyvidone collagen versus placebo, analyzing clinical improvement, biochemical response and quality of life in people over 60 years of age.

The Phase IV, double-blind, randomized, placebo-controlled clinical trial will be conducted between 2023 and 2026. Sixty patients with early-stage arthritis will participate, assessing factors such as pain, functionality and synovitis with various statistical tools and analyses.

DETAILED DESCRIPTION:
Geriatric rheumatology specializes in the study of rheumatic diseases in older adults, who have immune and physiological characteristics that influence the manifestation of these diseases. In the case of rheumatoid arthritis (RA), a chronic inflammatory disease that affects the joints, treatments that improve functionality and reduce pain in the hands, evaluated by ultrasound, are studied.

Its objective is to compare the effects of treatment with subcutaneous polyvidone collagen versus placebo on clinical improvement of the hands, biochemical response and quality of life in people over 60 years of age with rheumatoid arthritis.

A Phase IV, double-blind, randomized, placebo-controlled clinical trial will be conducted between August 2023 and August 2026. Sixty patients (30 in each group) with early-stage arthritis will participate. Pain, functionality, synovitis, and quality of life will be assessed using various scales, biochemical analyses, and statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with arthritic hand uni or bilateral
* Early rheumatoid arthritis (> or equal to 2 years of evolution with treatment and stable)
* Conventional treatment based on non-steroidal anti-inflammatory drugs (NSAIDs) alone for the disease without the use of biologic therapy or DMARDs.

Exclusion Criteria:

* Patient with previous treatment of the arthritic hand with steroids, previous surgery and/or some other local medical treatment
* Persistence of symptoms and functional alterations.
* Patients with diabetes mellitus, rheumatic polyarthropathy, scleroderma, fibromyalgia, systemic lupus erythematosus or any other autoimmune disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-07 (Actual)

PRIMARY OUTCOMES:
Effect of subcutaneous polyvidone collagen treatment on clinical hand recovery in adults with rheumatoid arthritis using the modified Kapandji Index, pain scale, and hand pressure strength. | Every 15 days for 2 months
  The clinical recovery of the hand in adults with rheumatoid arthritis will be evaluated by means of a modified Kapandji index, which consists of a test that allows evaluating the result of three different functions of the hand; the pain scale, where the patient is asked to observe the pain he/she feels and quantify it from 0 to 10, 0 being no pain and 10 being maximum pain; and the manual pressure force (MPF) where a maximum grip force is applied for a time of 3 seconds, with a rest of 1 minute between each repetition, making two attempts, measuring both times to obtain the best value.

SECONDARY OUTCOMES:
Effect of subcutaneous polyvidone collagen treatment in quality of life in adult rheumatoid arthritis | 2 months
  Quality of life will be assessed through the short SF-36 questionnaire. Applied at the time of the interview with each of the participants before and after the intervention in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes, 1, Principal Investigator — IMSS
Locations (2):
- Mexico (2):
  - National Western Speciality Hospital, Mexican Social Security Institute, Guadalajara, Jalisco
  - Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, México, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuzawa-Carballeda J, Alcocer-Varela J, Diaz de Leon L. Collagen-PVP decreases collagen turnover in synovial tissue cultures from rheumatoid arthritis patients. Ann N Y Acad Sci. 1999 Jun 30;878:598-602. doi: 10.1111/j.1749-6632.1999.tb07738.x. No abstract available. PMID 10415784
- [Background] Day AL, Curtis JR. Opioid use in rheumatoid arthritis: trends, efficacy, safety, and best practices. Curr Opin Rheumatol. 2019 May;31(3):264-270. doi: 10.1097/BOR.0000000000000602. PMID 30870218
- [Background] Safiri S, Kolahi AA, Hoy D, Smith E, Bettampadi D, Mansournia MA, Almasi-Hashiani A, Ashrafi-Asgarabad A, Moradi-Lakeh M, Qorbani M, Collins G, Woolf AD, March L, Cross M. Global, regional and national burden of rheumatoid arthritis 1990-2017: a systematic analysis of the Global Burden of Disease study 2017. Ann Rheum Dis. 2019 Nov;78(11):1463-1471. doi: 10.1136/annrheumdis-2019-215920. Epub 2019 Sep 11. PMID 31511227
- [Background] Alaya Z, Braham M, Aissa S, Kalboussi H, Bouajina E. A case of Caplan syndrome in a recently diagnosed patient with silicosis: A case report. Radiol Case Rep. 2018 Apr 11;13(3):663-666. doi: 10.1016/j.radcr.2018.03.004. eCollection 2018 Jun. PMID 30023036
- [Background] Curran AM, Naik P, Giles JT, Darrah E. PAD enzymes in rheumatoid arthritis: pathogenic effectors and autoimmune targets. Nat Rev Rheumatol. 2020 Jun;16(6):301-315. doi: 10.1038/s41584-020-0409-1. Epub 2020 Apr 27. PMID 32341463
- [Background] Scherer HU, Haupl T, Burmester GR. The etiology of rheumatoid arthritis. J Autoimmun. 2020 Jun;110:102400. doi: 10.1016/j.jaut.2019.102400. Epub 2020 Jan 22. PMID 31980337
- [Background] Damerau A, Gaber T. Modeling Rheumatoid Arthritis In Vitro: From Experimental Feasibility to Physiological Proximity. Int J Mol Sci. 2020 Oct 25;21(21):7916. doi: 10.3390/ijms21217916. PMID 33113770
- [Background] Aletaha D, Smolen JS. Diagnosis and Management of Rheumatoid Arthritis: A Review. JAMA. 2018 Oct 2;320(13):1360-1372. doi: 10.1001/jama.2018.13103. PMID 30285183
- [Background] Leon L, Abasolo L, Fernandez-Gutierrez B, Jover JA, Hernandez-Garcia C. Direct medical costs and their predictors in the EMAR-II cohort: "Variability in the management of rheumatoid arthritis and spondyloarthritis in Spain". Reumatol Clin (Engl Ed). 2018 Jan-Feb;14(1):4-8. doi: 10.1016/j.reuma.2016.09.006. Epub 2016 Oct 31. English, Spanish. PMID 27810462
- [Background] Kobak S, Bes C. An autumn tale: geriatric rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2018 Jan;10(1):3-11. doi: 10.1177/1759720X17740075. Epub 2017 Nov 7. PMID 29290762